CLINICAL TRIAL: NCT06852807
Title: Prospective Clinical Study of 18F-mFBG PET Imaging in Neuroblastoma
Brief Title: 18F-mFBG PET Imaging in the Evaluation of Neuroblastoma
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FAHZU-MFBG-NB
Record Dates: First submitted 2025-02-04; First posted 2025-02-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-01

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — 3-fluorobenzylguanidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-MFBG PET/CT in Neuroblastoma: Each patient receive a single intravenous injection of 18F-MFBG 2-5 MBq/kg and undergo PET/CT or PET/MR scan after 60 min post-injection.
  Interventions: Drug: 18F-MFBG

INTERVENTIONS:
Drug: 18F-MFBG — Patients with neuroblastoma malignancies receive 5.55 MBq/kg of 18F-MFBG intravenously followed by PET/CT or PET/MR after 60min of injection.

SUMMARY:
The aim of this study is to evaluate the diagnostic performance and tumor burden of 18F-metafluorobenzylguanidine (18F-MFBG) positron emission tomography (PET) in patients with neuroblastoma.

DETAILED DESCRIPTION:
Neuroblastoma highly expresses norepinephrine transporter (NET) which is targeted by function alanalogue of norepinephrine, 123/131I-MlBG. However, low spatial resolution of 123/131I-MlBG and inaccurate attenuation correction of single photon emission tomography (SPECT/CT) will affect the image quality of MlBG SPECT and lead to poor diagnosis of small lesions. In addition, 123l-MlBG imaging is usually performed at 24h after injection, while 131I-MlBG is performed at 48h or even 72h after injection. The procedure is complicated and takes a long time, which limits clinical application. 18F-labeled MFBG is an ideal tracer to show the expression of NET. Preliminary data show that 18F-MFBG imaging is safe and has favorable biodistribution and kinetics with good targeting of lesions. Patients can undergo PET 0.5 hours after injection without special preparation. Our study will assess the safety profile, image quality and evaluate the diagnostic performance and tumor burden of 18F-MFBG. Patients with suspected or histologically confirmed neuroblastoma will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-18 years old, with legal guardian;
2. Clinically suspected or confirmed patients with neuroblastoma;
3. If the patient is under 8 years old or unable to write, his/her guardian should understand and comply with the requirements of the study. If the patient is 8 years old or older and has written ability, both the patient and his/her guardian must sign the informed consent.

Exclusion Criteria:

1. Patients with severe primary diseases such as heart, brain, liver, kidney and hematopoietic system diseases;
2. Patients who have received ionizing radiation outside the scope of this experiment for other clinical medical or scientific research purposes within the past year, resulting in an annual radiation exposure dose exceeding 50 mSv.
3. Patients who have received experimental drugs or devices (with uncertain efficacy or safety) within one month;
4. Patients with any condition that the principal investigator of this study deems may cause harm or potential harm in any aspect related to this trial.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with suspected or confirmed neuroblastoma
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | through study completion, an average of 1.5 year
  Sensitivity, specificity, positive and negative predictive value of 18F-mFBG PET/CT and PET/MR Imaging in neuroblastoma

SECONDARY OUTCOMES:
18F-mFBG PET performence compared with other images | up to 24 months
  18F-mFBG PET performence compared with 18F-FDG PET or MRI, McNemar test, Two-tailed，P<.05
Prognostic Value of Baseline 18F-mFBG PET for Progression-Free Survival (PFS) in High-Risk Patients | through study completion, 3-4 years
  This measure evaluates the association between baseline 18F-mFBG PET parameters (e.g., SUVmax, SUVmean, metabolic tumor volume [MTV], total lesion glycolysis [TLG]) and progression-free survival (PFS) in high-risk neuroblastoma patients. PFS will be defined as the time from diagnosis to disease progression or relapse, assessed using the Kaplan-Meier method and Cox proportional hazards model.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China